CLINICAL TRIAL: NCT00705848
Title: Matrix Biology of Tracheobronchomalacia and Tracheal Stenosis
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Sidharta Gangadharan, Associate Professor of Surgery, Beth Israel Deaconess Medical Center
Other Study IDs: 2007P000336
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Tracheobronchomalacia; Tracheal Stenosis
Keywords: trachea; malacia; stenosis
MeSH Terms: conditions — Tracheobronchomalacia; Tracheal Stenosis; Tracheal Diseases; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Airway biopsies and brushings are to be used for staining and culture, respectively
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: 10 patients with tracheobronchomalacia
- 2: 10 patients with tracheal stenosis
- 3: 10 patients with normal airways (no known airway diseases)

SUMMARY:
It is not clearly understood what causes tracheobronchomalacia (weakening of the windpipe and airways) or tracheal stenosis (narrowing of the windpipe). We plan to take biopsies (small pieces of tissue) and brushings (to collect the cells that form the lining of the airway) from the airways of patients with these diseases and analyze these samples in a laboratory to try and determine the mechanism of disease. We will compare the results with that of patients with normal airways.

DETAILED DESCRIPTION:
* Controlled pilot study to determine whether there exists, at a molecular level, a predisposition to the development of tracheomalacia and subglottic stenosis. Thirty patients will be divided into 2 groups of 20 patients (study patients) and 10 patients (control group). Both groups will undergo bronchoscopy and airway biopsy
* The study is a pilot study to evaluate alterations in the airway matrix, growth factor levels, and vascular structures.in patients with tracheobronchomalacia and subglottic stenosis
* Bronchoscopies will be performed in the West Procedure UnitPulmonary Special Procedures Unit or in the operating room (depending on the clinical indication and patient scheduling) at the BIDMC after informed consent is obtained.
* Patients will receive topical upper airway anesthesia with lidocaine and intravenous conscious sedation with fentanyl and midazolam as per standard of care
* Biopsies will be performed according to standard protocols.
* Biopsies will be performed: 2 samples will be sent for pathology as part of clinical care and 2-3 samples used for research analysis.

ELIGIBILITY:
Inclusion Criteria:

* (study group): age ≥ 18, willingness and ability to give informed consent, clinical indication for bronchoscopy and biopsy, prior bronchoscopic diagnosis of tracheobronchomalacia, prior bronchoscopic diagnosis of subglottic stenosis (either idiopathic or post-intubation), and smoking cessation for ≥ 4 months. There is no gender or racial restriction. Pregnant women will not be included in the study because of the potential for hypoxemia (especially fetal) and prolongation of the procedure if complications arise. Patients must have family/friends to drive them home following the procedure.
* (control group): age ≥ 18, willingness and ability to give informed consent, clinical indication for bronchoscopy and biopsy, no prior diagnosis of any airway disease of any etiology, and smoking cessation for ≥ 4 months. There is no gender or racial restriction. Pregnant women will not be included in the study because of the potential for hypoxemia (especially fetal) and prolongation of the procedure if complications arise. Patients must have family/friends to drive them home following the procedure.

Exclusion Criteria:

* (study group): pre-existing airway disorders other than tracheobronchomalacia or subglottic stenosis, etiology of subglottic stenosis other than idiopathic or post-intubation, pulmonary vascular disease, inability to tolerate intravenous conscious sedation.
* (control group): any pre-existing airway disorder, pulmonary vascular disease, and inability to tolerate intravenous conscious sedation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with tracheobronchomalacia or tracheal stenosis referred to this tertiary care facility
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2008-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sidhu Gangadharan, M.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No